CLINICAL TRIAL: NCT02801409
Title: Effects of Epidural Anesthesia-analgesia on Long-term Survival in Patients After Lung Cancer Surgery: A Randomized Controlled Trial
Brief Title: Epidural Anesthesia-analgesia and Long-term Survival After Lung Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2013[653]; ChiCTR-TRC-14004136 (Registry Identifier: Chinese Clinical Trial Registry (www.chictr.org.cn))
Record Dates: First submitted 2016-06-12; First posted 2016-06-15 (Estimated); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Lung Cancer; Thoracic Surgery; Anesthesia, Epidural; Neoplasm Recurrence, Local; Neoplasm Metastasis
Keywords: Lung Cancer; Surgical Resection; Epidural Anesthesia and Analgesia; Cancer recurrence/metastasis; Long-Term Outcome
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Recurrence, Local; Neoplasm Metastasis; Agnosia | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia alone (Active Comparator): General anesthesia is performed during surgery; patient-controlled intravenous analgesia is provided after surgery.
  Interventions: Drug: General anesthesia alone
- Combined epidural-general anesthesia (Experimental): Combined epidural-general anesthesia is performed during surgery; patient-controlled epidural analgesia is provided after surgery.
  Interventions: Drug: Combined epidural-general anesthesia

INTERVENTIONS:
Drug: General anesthesia alone — General anesthesia is performed during surgery; patient-controlled intravenous analgesia is provided after surgery.
  Arms: General anesthesia alone
Drug: Combined epidural-general anesthesia — Combined epidural-general anesthesia is performed during surgery; patient-controlled epidural analgesia is provided after surgery.
  Arms: Combined epidural-general anesthesia

SUMMARY:
Available studies suggest that regional anesthesia-analgesia may decrease the occurrence of recurrence/metastasis in patients after cancer surgery. However, evidences from prospective studies are still lacking. The purpose of this randomized controlled trial is to investigate the effect of epidural anesthesia-analgesia on recurrence-free survival in patients undergoing lung cancer surgery.

DETAILED DESCRIPTION:
Lung cancer is increasing and is the leading cause of cancer death. Surgical resection is the mainstay of treatment for early stage non-small cell lung cancer. However, long-term survival after lung cancer surgery is far from optimal, and cancer recurrence or metastasis is the main reason leading to cancer death in these patients.

The development of cancer recurrence/metastasis largely depends on the balance between tumor-promoting factors and immune function of the body. Studies showed that surgical manipulation releases cancer cells into circulation; and stress response induced by surgery inhibits the cell-mediated immunity. In addition, volatile anesthetics and opioids may also aggravate immunosuppression and potentially worsen long-term outcome. On the other hand, regional anesthesia can blunt surgical stress and reduce anesthetic consumption. These effects may help to preserve immune function and reduce recurrence/metastasis. However, existing evidences are insufficient to draw conclusion in this topic.

The purpose of this randomized controlled trial is to test the hypothesize that regional anesthesia-analgesia may reduce recurrence/metastasis and improve long-term survival in patients after lung cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (aged 18-80 years);
2. Clinically diagnosed as primary non-small cell lung cancer of stage IA to IIIA, and scheduled for radical surgery;
3. Agreed to receive patient-controlled analgesia after surgery.

Exclusion Criteria:

1. Distant metastasis, malignant tumor in other organs, or chemo-/radiotherapy or other anti-cancer therapy before surgery;
2. Comorbid with autoimmune diseases, or glucocorticoid/immunosuppressant therapy within 1 year;
3. History of schizophrenia, epilepsy or Parkinson disease, or unable to complete preoperative assessment due to severe dementia, language barrier, or end-stage disease;
4. Severe hepatic disease (Child-Pugh classification C), renal failure (serum creatinine >442 umol/L or receiving renal replacement therapy), or American Society of Anesthesiologists classification IV or higher;
5. History of anesthesia and/or surgery within 1 year;
6. Contraindications to epidural anesthesia, including spinal deformity, coagulation dysfunction, local infection, and history of spinal trauma/surgery;
7. Allergic to any medications used during the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2015-05-25 (Actual); Primary Completion 2017-11-11 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survival after surgery. | Up to 4 years after surgery.
  Time from surgery to the earliest date of recurrence/metastasis or death from any cause, whichever came first.

SECONDARY OUTCOMES:
Rate of intensive care unit admission after surgery. | Up to 30 days after surgery.
  Rate of intensive care unit admission after surgery.
Incidence of postoperative complications during hospital stay. | Up to 30 days after surgery.
  Postoperative complications are defined as new-onset conditions that are harmful to patients' recovery and required therapeutic intervention, i.e., class II or higher on the Clavien-Dindo classification.
Duration of chest tube placement. | Up to 30 days after surgery.
  Duration of chest tube placement.
Length of stay in hospital after surgery. | Up to 30 days after surgery.
  Length of stay in hospital after surgery.
Rate of all-cause mortality during hospital stay after surgery. | Up to 30 days after surgery.
  Rate of all-cause mortality during hospital stay after surgery.
Overall survival rate after surgery. | Up to 4 year after surgery.
  Time from surgery to all-cause death.
Cancer-specific survival after surgery. | Up to 4 years after surgery.
  Time from surgery to cancer-specific death; deaths from other causes are censored at the time of death.
Activity engagement in 1-year survivors. | At the end of the first year after surgery.
  Activity engagement is assessed by estimating metabolic equivalents (METs; 1 MET = 3·5 ml/min/kg resting oxygen consumption) for activity in daily life.

OTHER OUTCOMES:
Pain intensity after surgery. | During the first 3 days after surgery.
  Assessed with the numeric rating score, an 11-point scale where 0 = no pain and 10 = the most severe pain.
Recurrence-free survival in cancer patients. | Up to 4 years after surgery.
  Time from surgery to the earliest date of recurrence/metastasis or death from any cause, whichever came first.
Overall survival in cancer patients. | Up to 4 years after surgery.
  Time from surgery to all-cause death.
Cancer-specific survival in cancer patients. | Up to 4 years after surgery.
  Time from surgery to cancer-specific death; deaths from other causes are censored at the time of death.
Number of CD8+ and FOXP3+ T cells per mm2 tumor area (sub-study). | After resection of lung adenocarcinoma specimens
  Immunohistochemical staining of CD8 and FOXP3 molecules in excised lung adenocarcinoma specimens. Performed in part of enrolled patients.
Percentage of NK-cells and T-cell subgroups in peripheral blood (sub-study). | Peripheral blood samples collected before induction, at the end of surgery and at 24 hours after surgery.
  Measured by flow cytometry. Performed in part of enrolled patients.
Rate of chronic pain at 3 month and 6 month after surgery (sub-study). | At 3 months and 6 months after surgery.
  Chronic pain is measured with the Brief Pain Inventory (BPI), neuropathic pain screening questionnaire (ID pain), and McGill Pain Questionnair (MPQ). Performed in part of enrolled patients.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelsey CR, Marks LB, Hollis D, Hubbs JL, Ready NE, D'Amico TA, Boyd JA. Local recurrence after surgery for early stage lung cancer: an 11-year experience with 975 patients. Cancer. 2009 Nov 15;115(22):5218-27. doi: 10.1002/cncr.24625. PMID 19672942
- [Background] Sawyer TE, Bonner JA, Gould PM, Foote RL, Deschamps C, Lange CM, Li H. Factors predicting patterns of recurrence after resection of N1 non-small cell lung carcinoma. Ann Thorac Surg. 1999 Oct;68(4):1171-6. doi: 10.1016/s0003-4975(99)00678-5. PMID 10543475
- [Background] Snyder GL, Greenberg S. Effect of anaesthetic technique and other perioperative factors on cancer recurrence. Br J Anaesth. 2010 Aug;105(2):106-15. doi: 10.1093/bja/aeq164. PMID 20627881
- [Background] Koebel CM, Vermi W, Swann JB, Zerafa N, Rodig SJ, Old LJ, Smyth MJ, Schreiber RD. Adaptive immunity maintains occult cancer in an equilibrium state. Nature. 2007 Dec 6;450(7171):903-7. doi: 10.1038/nature06309. Epub 2007 Nov 18. PMID 18026089
- [Background] Shakhar G, Ben-Eliyahu S. Potential prophylactic measures against postoperative immunosuppression: could they reduce recurrence rates in oncological patients? Ann Surg Oncol. 2003 Oct;10(8):972-92. doi: 10.1245/aso.2003.02.007. PMID 14527919
- [Background] Yamaguchi K, Takagi Y, Aoki S, Futamura M, Saji S. Significant detection of circulating cancer cells in the blood by reverse transcriptase-polymerase chain reaction during colorectal cancer resection. Ann Surg. 2000 Jul;232(1):58-65. doi: 10.1097/00000658-200007000-00009. PMID 10862196
- [Background] Hofer SO, Molema G, Hermens RA, Wanebo HJ, Reichner JS, Hoekstra HJ. The effect of surgical wounding on tumour development. Eur J Surg Oncol. 1999 Jun;25(3):231-43. doi: 10.1053/ejso.1998.0634. PMID 10336800
- [Background] Lennard TW, Shenton BK, Borzotta A, Donnelly PK, White M, Gerrie LM, Proud G, Taylor RM. The influence of surgical operations on components of the human immune system. Br J Surg. 1985 Oct;72(10):771-6. doi: 10.1002/bjs.1800721002. PMID 2412626
- [Background] Carter JJ, Whelan RL. The immunologic consequences of laparoscopy in oncology. Surg Oncol Clin N Am. 2001 Jul;10(3):655-77. PMID 11685934
- [Background] Tashiro T, Yamamori H, Takagi K, Hayashi N, Furukawa K, Nitta H, Toyoda Y, Sano W, Itabashi T, Nishiya K, Hirano J, Nakajima N. Changes in immune function following surgery for esophageal carcinoma. Nutrition. 1999 Oct;15(10):760-6. doi: 10.1016/s0899-9007(99)00151-3. PMID 10501289
- [Background] Downing JE, Miyan JA. Neural immunoregulation: emerging roles for nerves in immune homeostasis and disease. Immunol Today. 2000 Jun;21(6):281-9. doi: 10.1016/s0167-5699(00)01635-2. PMID 10825740
- [Background] Elenkov IJ, Wilder RL, Chrousos GP, Vizi ES. The sympathetic nerve--an integrative interface between two supersystems: the brain and the immune system. Pharmacol Rev. 2000 Dec;52(4):595-638. PMID 11121511
- [Background] Page GG, Blakely WP, Ben-Eliyahu S. Evidence that postoperative pain is a mediator of the tumor-promoting effects of surgery in rats. Pain. 2001 Feb 1;90(1-2):191-9. doi: 10.1016/s0304-3959(00)00403-6. PMID 11166986
- [Background] Afsharimani B, Cabot PJ, Parat MO. Morphine use in cancer surgery. Front Pharmacol. 2011 Aug 8;2:46. doi: 10.3389/fphar.2011.00046. eCollection 2011. PMID 21852973
- [Background] Xu YX, Ayala A, Chaudry IH. Prolonged immunodepression after trauma and hemorrhagic shock. J Trauma. 1998 Feb;44(2):335-41. doi: 10.1097/00005373-199802000-00018. PMID 9498507
- [Background] Klein HG. Immunomodulatory aspects of transfusion: a once and future risk? Anesthesiology. 1999 Sep;91(3):861-5. doi: 10.1097/00000542-199909000-00040. No abstract available. PMID 10485799
- [Background] Gottschalk A, Sharma S, Ford J, Durieux ME, Tiouririne M. Review article: the role of the perioperative period in recurrence after cancer surgery. Anesth Analg. 2010 Jun 1;110(6):1636-43. doi: 10.1213/ANE.0b013e3181de0ab6. Epub 2010 Apr 30. PMID 20435944
- [Background] Ishihara Y, Matsunaga K, Iijima H, Fujii T, Oguchi Y, Kagawa J. Time-dependent effects of stressor application on metastasis of tumor cells in the lung and its regulation by an immunomodulator in mice. Psychoneuroendocrinology. 1999 Oct;24(7):713-26. doi: 10.1016/s0306-4530(99)00023-2. PMID 10451907
- [Background] Freire-Garabal M, Nunez MJ, Balboa JL, Fernandez-Rial JC, Vallejo LG, Gonzalez-Bahillo J, Rey-Mendez M. Effects of alprazolam on cellular immune response to surgical stress in mice. Cancer Lett. 1993 Sep 30;73(2-3):155-60. doi: 10.1016/0304-3835(93)90258-b. PMID 8221628
- [Background] Andersen BL, Farrar WB, Golden-Kreutz D, Kutz LA, MacCallum R, Courtney ME, Glaser R. Stress and immune responses after surgical treatment for regional breast cancer. J Natl Cancer Inst. 1998 Jan 7;90(1):30-6. doi: 10.1093/jnci/90.1.30. PMID 9428780
- [Background] Heaney A, Buggy DJ. Can anaesthetic and analgesic techniques affect cancer recurrence or metastasis? Br J Anaesth. 2012 Dec;109 Suppl 1:i17-i28. doi: 10.1093/bja/aes421. PMID 23242747
- [Background] Conrick-Martin I, Buggy DJ. The effects of anesthetic and analgesic techniques on immune function. J Clin Anesth. 2013 Jun;25(4):253-4. doi: 10.1016/j.jclinane.2013.04.003. Epub 2013 Apr 26. No abstract available. PMID 23624071
- [Background] Ahlers O, Nachtigall I, Lenze J, Goldmann A, Schulte E, Hohne C, Fritz G, Keh D. Intraoperative thoracic epidural anaesthesia attenuates stress-induced immunosuppression in patients undergoing major abdominal surgery. Br J Anaesth. 2008 Dec;101(6):781-7. doi: 10.1093/bja/aen287. Epub 2008 Oct 15. PMID 18922851
- [Background] Piegeler T, Votta-Velis EG, Liu G, Place AT, Schwartz DE, Beck-Schimmer B, Minshall RD, Borgeat A. Antimetastatic potential of amide-linked local anesthetics: inhibition of lung adenocarcinoma cell migration and inflammatory Src signaling independent of sodium channel blockade. Anesthesiology. 2012 Sep;117(3):548-59. doi: 10.1097/ALN.0b013e3182661977. PMID 22846676
- [Background] Waurick R, Van Aken H. Update in thoracic epidural anaesthesia. Best Pract Res Clin Anaesthesiol. 2005 Jun;19(2):201-13. doi: 10.1016/j.bpa.2004.12.001. PMID 15966493
- [Background] Biki B, Mascha E, Moriarty DC, Fitzpatrick JM, Sessler DI, Buggy DJ. Anesthetic technique for radical prostatectomy surgery affects cancer recurrence: a retrospective analysis. Anesthesiology. 2008 Aug;109(2):180-7. doi: 10.1097/ALN.0b013e31817f5b73. PMID 18648226
- [Background] Exadaktylos AK, Buggy DJ, Moriarty DC, Mascha E, Sessler DI. Can anesthetic technique for primary breast cancer surgery affect recurrence or metastasis? Anesthesiology. 2006 Oct;105(4):660-4. doi: 10.1097/00000542-200610000-00008. PMID 17006061
- [Background] Tsui BC, Rashiq S, Schopflocher D, Murtha A, Broemling S, Pillay J, Finucane BT. Epidural anesthesia and cancer recurrence rates after radical prostatectomy. Can J Anaesth. 2010 Feb;57(2):107-12. doi: 10.1007/s12630-009-9214-7. PMID 19911247
- [Background] Lin L, Liu C, Tan H, Ouyang H, Zhang Y, Zeng W. Anaesthetic technique may affect prognosis for ovarian serous adenocarcinoma: a retrospective analysis. Br J Anaesth. 2011 Jun;106(6):814-22. doi: 10.1093/bja/aer055. Epub 2011 Mar 24. PMID 21436156
- [Background] Cummings KC 3rd, Xu F, Cummings LC, Cooper GS. A comparison of epidural analgesia and traditional pain management effects on survival and cancer recurrence after colectomy: a population-based study. Anesthesiology. 2012 Apr;116(4):797-806. doi: 10.1097/ALN.0b013e31824674f6. PMID 22273991
- [Background] Ismail H, Ho KM, Narayan K, Kondalsamy-Chennakesavan S. Effect of neuraxial anaesthesia on tumour progression in cervical cancer patients treated with brachytherapy: a retrospective cohort study. Br J Anaesth. 2010 Aug;105(2):145-9. doi: 10.1093/bja/aeq156. Epub 2010 Jun 23. PMID 20573631
- [Background] Lai R, Peng Z, Chen D, Wang X, Xing W, Zeng W, Chen M. The effects of anesthetic technique on cancer recurrence in percutaneous radiofrequency ablation of small hepatocellular carcinoma. Anesth Analg. 2012 Feb;114(2):290-6. doi: 10.1213/ANE.0b013e318239c2e3. Epub 2011 Nov 21. PMID 22104077
- [Background] Gupta A, Bjornsson A, Fredriksson M, Hallbook O, Eintrei C. Reduction in mortality after epidural anaesthesia and analgesia in patients undergoing rectal but not colonic cancer surgery: a retrospective analysis of data from 655 patients in central Sweden. Br J Anaesth. 2011 Aug;107(2):164-70. doi: 10.1093/bja/aer100. Epub 2011 May 17. PMID 21586443
- [Background] Christopherson R, James KE, Tableman M, Marshall P, Johnson FE. Long-term survival after colon cancer surgery: a variation associated with choice of anesthesia. Anesth Analg. 2008 Jul;107(1):325-32. doi: 10.1213/ane.0b013e3181770f55. PMID 18635504
- [Background] Gottschalk A, Ford JG, Regelin CC, You J, Mascha EJ, Sessler DI, Durieux ME, Nemergut EC. Association between epidural analgesia and cancer recurrence after colorectal cancer surgery. Anesthesiology. 2010 Jul;113(1):27-34. doi: 10.1097/ALN.0b013e3181de6d0d. PMID 20508494
- [Background] Wuethrich PY, Hsu Schmitz SF, Kessler TM, Thalmann GN, Studer UE, Stueber F, Burkhard FC. Potential influence of the anesthetic technique used during open radical prostatectomy on prostate cancer-related outcome: a retrospective study. Anesthesiology. 2010 Sep;113(3):570-6. doi: 10.1097/ALN.0b013e3181e4f6ec. PMID 20683253
- [Background] Myles PS, Peyton P, Silbert B, Hunt J, Rigg JR, Sessler DI; ANZCA Trials Group Investigators. Perioperative epidural analgesia for major abdominal surgery for cancer and recurrence-free survival: randomised trial. BMJ. 2011 Mar 29;342:d1491. doi: 10.1136/bmj.d1491. PMID 21447587
- [Background] Taylor MD, Nagji AS, Bhamidipati CM, Theodosakis N, Kozower BD, Lau CL, Jones DR. Tumor recurrence after complete resection for non-small cell lung cancer. Ann Thorac Surg. 2012 Jun;93(6):1813-20; discussion 1820-1. doi: 10.1016/j.athoracsur.2012.03.031. Epub 2012 Apr 26. PMID 22542070
- [Background] Alberts WM. Follow up and surveillance of the patient with lung cancer: what do you do after surgery? Respirology. 2007 Jan;12(1):16-21. doi: 10.1111/j.1440-1843.2006.00956.x. PMID 17207020
- [Background] Colt HG, Murgu SD, Korst RJ, Slatore CG, Unger M, Quadrelli S. Follow-up and surveillance of the patient with lung cancer after curative-intent therapy: Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):e437S-e454S. doi: 10.1378/chest.12-2365. PMID 23649451
- [Background] Bruzzi JF, Munden RF. PET/CT imaging of lung cancer. J Thorac Imaging. 2006 May;21(2):123-36. doi: 10.1097/00005382-200605000-00004. PMID 16770229
- [Background] Pei L, Tan G, Wang L, Guo W, Xiao B, Gao X, Wang L, Li H, Xu Z, Zhang X, Zhao J, Yi J, Huang Y. Comparison of combined general-epidural anesthesia with general anesthesia effects on survival and cancer recurrence: a meta-analysis of retrospective and prospective studies. PLoS One. 2014 Dec 30;9(12):e114667. doi: 10.1371/journal.pone.0114667. eCollection 2014. PMID 25548913